CLINICAL TRIAL: NCT00705185
Title: Exploring Potential Serum/Plasma-Based Biomarkers as a Test for Major Depressive Disorder Diagnostics ("Bio-Test MDD")
Brief Title: Exploring a Potential Blood Test to Diagnose Major Depressive Disorder
Acronym: Bio-TestMDD
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Precision Human Biolaboratories (Unknown); Cambridge Health Alliance (Other); University of Connecticut (Other); Vanderbilt University (Other); Psychiatric Medicine Associates, L.L.C. (Other)
Responsible Party: George I. Papakostas, M.D., Massachusetts General Hospital
Other Study IDs: 2007-P-002525
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Blood Test
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Adults with Major Depressive Disorder- as defined by the criteria in the DSM-IV
- 2: Healthy Controls- research subjects who have not met criteria for any lifetime Axis-I disorder (DSM-IV)

SUMMARY:
The purpose of this study is to develop a blood test for major depression and measure the effects of ziprasidone monotherapy on these markers.

Specific Aim: Using a multiplex biomarker assay we will measure levels of 16 biomarkers in patients with MDD enrolled in this ancillary study (adjunct to study NCT00555997) and compare these results to those of healthy controls" (defined as research subjects who have not met criteria for any lifetime Axis-I disorder (DSM-IV)) from an existing dataset at PHB.

DETAILED DESCRIPTION:
This proposed study will be an ancillary study to clinical trial NCT00555997 (www.clinicaltrials.gov) entitled: "A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Sequential Trial of Ziprasidone as Monotherapy for Major Depressive Disorder" (MDD)." Precision Human Biolaboratory ("PHB") is attempting to develop a proprietary blood test intended to potentially serve as a biological marker ("bio-marker") for MDD. Specifically, PHB's research team will employ a unique approach towards developing a diagnostic test for MDD: measures from multiple blood-based biological markers will be obtained from patients with MDD and then analyzed with the use of several interrelated algorithms in order to derive a single biological measure ("bio-marker") with a high predictive value for MDD. PHBs' test panel of blood-based biological markers will consist of a number of cytokines, stress related hormones, and binding proteins that have each been linked to MDD. This innovative test panel is expected to provide general practice physicians with a tool to more accurately identify and classify patients with MDD which, in turn, could potentially , allow for the more effective monitoring of pharmacotherapy (antidepressant drug therapy). Thus, the development of a highly reliable biomarker for MDD could improve the standard of care for depression.

For this ancillary study, 120 antidepressant-free outpatients with MDD who have been deemed eligible to participate in trial NCT00555997 will be recruited from participating centers. Participating subjects will undergo a blood draw during the baseline visit for NCT00555997. Values obtained will be compared with those of "healthy controls" (defined as research subjects who have not met criteria for any lifetime Axis-I disorder (DSM-IV)) from an existing dataset at PHB.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65.

* Written informed consent.
* MDD, current according to the fourth version of the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV) as diagnosed by the Mini International Neuropsychiatric Interview (MINI; Sheehan et al, 1998).
* Quick Inventory of Depressive Symptomatology - Self-Rated (QIDS-SR- Trivedi et al, 2004) score of at least 10 at both screen and baseline visits.

Exclusion Criteria:

* Pregnant women.
* Women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or a partner with vasectomy).
* Treatment with antidepressants for 2 weeks prior to the screen visit. If interested in discontinuing their current medication, potential participants must discuss this possibility with the prescribing physician. Study doctors will not implement any form of treatment washout.
* Patients who no longer meet DSM-IV criteria for MDD during the baseline visit, or patients who demonstrate a 25% or greater reduction in QIDS-SR scores, screening to baseline.
* Serious suicide or homicide risk, as assessed by the evaluating clinician or a score of 4 on the third item of the HAM-D.
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
* Patients who meet criteria for alcohol or substance dependence, active within the last month.
* Any bipolar disorder (current or past).
* Any psychotic disorder (current or past).
* Psychotic features in the current episode or a history of psychotic features.
* History of a seizure disorder.
* Clinical or laboratory evidence of untreated hypothyroidism.
* Patients requiring excluded medications (see table 1 for details).
* Prior course of ziprasidone, or intolerance to ziprasidone at any dose.
* Any investigational psychotropic drug within the last 3 months.
* Patients with significant cardiac conduction problems on screening electrocardiogram such as atrial fibrillation, atrial flutter, atrio-ventricular block, prolonged or abnormal QTc interval (i.e. QTc>450msec), or prolonged QRS interval.
* Patients who have suffered a myocardial infarction within the past 12 months, with uncompensated heart failure, or a history of QTc prolongation.
* Patients with abnormal serum potassium or magnesium levels upon screening.
* Patients currently taking other drugs that prolong the QTc including dofetilide, sotalol, quinidine, class Ia antiarrhythmics, class III antiarrhythmics, mesoridazine, thioridazine, chlorpromazine, droperidol, pimozide, sparfloxacin, gatifloxacin, moxifloxacin, halofantrine, mefloquine, pentamidine, arsenic trioxide, levomethadyl acetate, dolasetron methylate, probucol or tacrolimus.
* Patients who have failed to experience significant clinical improvement following 3 or more antidepressant trials of adequate duration (at least 6 weeks) and dose (minimal effective doses defined as: fluoxetine, paroxetine, citalopram 20mg; sertraline, fluvoxamine 50mg, escitalopram 10mg, paroxetine CR 25mg, venlafaxine 75mg, duloxetine 60mg, bupropion 150mg, 15mg of mirtazapine, trazodone or nefazodone 300mg).
* The presence of Addison's or Cushing's disease.
* The presence of rheumatoid arthritis, or systemic lupus erythematosus.
* The regular use of non-steroidal anti-inflammatory medications or oral steroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Major Depressive Disorder (DSM-IV)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
16 Biological Markers; Group comparison between adults with Major Depressive Disorder and healthy controls | Screen visit

CONTACTS AND LOCATIONS:
Overall Officials: George I Papakostas, M.D., Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Psychiatric Medicine Associates, L.L.C., Chicago, Illinois
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee